CLINICAL TRIAL: NCT07155941
Title: Ecological Momentary Intervention for Reward in Anhedonia
Acronym: EMIRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMIRA
Record Dates: First submitted 2025-07-30; First posted 2025-09-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Anhedonia; Anxiety; Stress; Depression
MeSH Terms: conditions — Anhedonia; Anxiety Disorders; Depression | interventions — Sensitivity and Specificity; Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reward Training (Experimental)
  Interventions: Behavioral: Training of reward processing/sensitivity; Other: Psychoeducation
- Relaxation Training (Active Comparator)
  Interventions: Behavioral: Relaxation Training (PMR); Other: Psychoeducation

INTERVENTIONS:
Behavioral: Training of reward processing/sensitivity — Participants in the experimental group complete a two-week ecological momentary intervention (EMI) consisting of three brief training units per day, each delivered via a smartphone. The exercises target different aspects of reward processing and are scheduled at specific times throughout the day.
  The morning unit (to be completed between 10:00 and 12:00 a.m.) involves a positive mental imagery task guided by audio recording. Participants are guided to vividly imagine a future situation with the most pleasurable and meaningful outcome possible. They are encouraged to mentally activate all senses, thoughts, and emotions associated with this scenario.
  The afternoon unit (to be completed between 3:00 and 5:00 p.m.) consists of a savoring exercise guided by audio recording. Participants recall a positive experience from the past and are instructed to re-experience and savor it mentally by focusing on its sensory details, emotional quality, and personal significance.
  The evening unit (to be
  Arms: Reward Training
Behavioral: Relaxation Training (PMR) — Participants in the control group complete a two-week progressive muscle relaxation (PMR) program designed to match the reward training in both frequency and duration. The intervention consists of three daily units, each delivered via a smartphone app and guided by audio recordings.
  The first and second units of each day consist of short audio-guided PMR sessions (approximately 5 minutes each). These exercises systematically guide participants through alternating tension and relaxation of different muscle groups to promote physical and mental relaxation.
  The third unit of the day focuses on reflection. Participants are asked to evaluate their experiences with the relaxation exercises over the course of the day. They reflect on their ability to engage with the exercises, the perceived effects (e.g., feelings of relaxation), any difficulties they encountered, and strategies to enhance the effectiveness of relaxation in their daily life beyond the intervention.
  Arms: Relaxation Training
Other: Psychoeducation — All participants receive a psychoeducation session on the day before the respective intervention starts. In this session, a graduate-level study team member introduces the rationale behind the training (PMR or reward-training), and demonstrates each exercise. Participants also practice each task.

SUMMARY:
The present study evaluates a two week ecological momentary intervention (EMI) in reducing anhedonia and psychological distress (i.e. elevated depression, stress and anxiety). Participants in the experimental group complete three daily exercises targeting reward-related processes, including positive mental imagery, savoring, gratitude, taking ownership for positive experience, and silver lining. These components were selected to improve reward anticipation as well as reward consumption and reward learning as the underlying mechanisms of anhedonia. An active control group receives progressive muscle relaxation training, matched in format and frequency. Exercise units are presented using audio recordings via smartphone app.

DETAILED DESCRIPTION:
Anhedonia, the diminished ability to experience positive emotions such as pleasure, is a clinically relevant condition central to depression and frequently observed across a range of other psychological disorders including anxiety disorders or chronic stress. Despite its prevalence and impact on quality of life, effective interventions specifically targeting anhedonia remain limited. Standard cognitive-behavioral therapies (CBT) often reduce negative affect (e.g., sadness, anxiety) but tend to be less effective in enhancing positive affect. Moreover, anhedonia has been proposed as a potential limiting factor in the efficacy of exposure-based treatments for anxiety disorders, underscoring the need for low-threshold interventions that directly target reward-related deficits.

At the core of anhedonia lies impaired reward processing, which involves multiple phases: (1) reward anticipation (wanting), (2) reward consumption (liking), and (3) reward-based learning. Individuals with elevated anhedonia often show deficits across these domains, leading to reduced engagement in rewarding activities and motivational impairments. Therefore, effective interventions should aim to strengthen these specific facets of reward functioning.

Emerging approaches such as Positive Affect Treatment (PAT) have demonstrated promising effects by combining components like positive mental imagery, savoring, self-reinforcement (i.e., taking ownership of positive experiences), and cognitive reframing (e.g., silver lining techniques). Complementary evidence suggests that gratitude-based interventions can enhance well-being and buffer against stress, based on the idea that gratitude and negative affect are partially incompatible.

Building on these findings, the current study tests a two-week ecological momentary intervention (EMI) designed to enhance reward processing and reduce anhedonia in daily life. The intervention is delivered via the smartphone app m-Path and comprises three brief training units per day. These include a combination of audio-guided exercises and ecological momentary assessments (EMA) capturing mood, activity, and psychological symptoms. The exercises target positive mental imagery, savoring, gratitude, silver lining, and taking ownership of positive experiences-each mapped onto distinct components of reward processing. EMI formats offer the advantage of flexibility and integration into everyday contexts without requiring direct clinician contact.

Participants are randomly assigned to either the reward-focused intervention group or an active control group. The control group receives a structurally equivalent two-week training consisting of progressive muscle relaxation (PMR) exercises, also delivered via the m-Path app. PMR is an established stress-reduction technique and serves as an active comparator matched in format, frequency, and duration. The control group completes two audio-guided PMR sessions per day and one brief reflection unit each evening.

It is hypothesized that the reward intervention will (a) reduce anhedonia and psychological distress more effectively than PMR and (b) lead to specific improvements in reward processing.

ELIGIBILITY:
Inclusion Criteria:

* German speaking
* Smartphone available and willingness to participate in repeated training units and questions delivered via app
* Clinically elevated anhedonia (SHAPS >= 25) and elevated depression (DASS-21-Depression >= 10), elevated anxiey (DASS-21-Anxiety >= 6) or elevated stress (DASS-21-Stress >= 10)

Exclusion Criteria:

* Psychotropic medication
* Psychotherapy currently ongoing or planned during participation
* Suicidality, lifetime diagnosis of bipolar disorders or psychotic episodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in anhedonia/hedonic capacity; measured with the Snaith-Hamilton Pleasure Scale (SHAPS) from baseline to post-intervention and baseline to 3-months follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale consists of 14 items rated on a four-point Likert-scale (1 = "I completely agree", 2 = "I agree", 3 = "I do not agree", 4 = "I completely disagree"). The SHAPS assesses participants' hedonic capacity/ability to feel pleasure. Sum scores range from 14 to 56, with a higher scores indicating more pronounced anhedonia. The scale is a standard survey method for anhedonia and has been validated by a large number of studies.
Change in depression, anxiety and stress; measured with the Depression-Anxiety-Stress-Scale (DASS-21) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The questionnaire consists of 21 items rated on a four-point Likert-scale (0 = "Didn't apply to me at all", 1 = "Applied to me to a certain extent or sometimes", 2 = "Applied to me to a considerable extent or quite often", 3 = "Applied very strongly to me, or most of the time"). The questionnaire is used to assess the severity of depressive, and anxiety symptoms as well as symptoms of distress during the last week. Scores range from 0 to 63 with the overall score being an indicator of general psychopathology. Subscales for depression, anxiety and stress exist. The scale is a widely used survey method and has proven to be a valid measure many times.

SECONDARY OUTCOMES:
Change in anhedonia; measured with the Dimensional Anhedonia Rating Scale (DARS) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The DARS is a 26-item scale (every item 5-point with 0 = "not at all", 1 = "a little", 2 = "moderately", 3 = "mostly", 4 = "very") that can be used to assess anhedonia/ability to respond to reward. Its advantage is that the subjects can rate their ability to enjoy certain activities/areas of reinforcement (non-social positive activities, favourite foods/drinks, positive social activities and sensory experiences) using their own examples and thus increased validity. Its value range extends from 0 to 104 with high values indicating higher reward responsiveness and thus lower anhedonia.
Change in reward sensitivity and procession; measured with the Positive Valence System Scale-21 (PVSS-21) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale consists of 21 9-point-items (1 = "extremely unapplicable", 5 = "neutral", 9 = "extremely applicable" to assess one's ability to process reward/the systems of positive valence (Reward valuation, reward expectancy, effort valuation, reward anticipation, initial responsiveness and reward satiation) as introduced by the NIMH-Research Domain Criteria using different areas of reward as examples (food, physical touch, outdoors, positive feedback, social interactions, hobbies and goals). Its value range extends from 21 to 189 with higher values indicating more pronounced reward processing abilities.
Trait-Positive Emotionality (PE) and its change as measured with the NEO-Five-Factor (NEO-FFI) Positive-Emotionality-Subscale from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale consists of four five-point items (1 = "strong rejection", 2 = "rejection", 3 = "neutral", 4 = "approval", 5 = "strong approval") with a value range extending from 4 to 20. Second and fourth item are reverse coded. Higher values indicating higher ability to experience positive emotions easily.
Positive and negative affect and their changes; measured with the Positive and Negative Affect Schedule (PANAS) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The PANAS consists of two 10-items scales, one measuring Positive Affect (PA) and the other measuring Negative Affect (NA). Each item on the measure is rated on a 5-point scale (1=not at all; 2=a little; 3=moderately; 4= quite a bit; and 5=extremely). Positive Affect (PA) "reflects the extent to which a person feels enthusiastic, active, and alert". Negative Affect (NA) is a "general dimension of subjective distress and unpleasurable engagement that subsumes a variety of aversive mood states". Higher scores on the PA dimension indicate a greater extent of positive affect, higher scores on the NA dimension indicate a greater extent of negative affect.
Change in social anxiety; measured with the Social Phobia Inventory (SPIN) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The SPIN is a widely used and well-validated questionnaire to assess social anxiety. It presents a general assessment of social anxiety symptoms and consists of 17 four-point items (1 = "not stressed at all", 2 = "lightly stressed", 3 = "quite stressed", 4 = "heavily stressed", 5 = "extremely stressed") with a value range extending from 17 to 68; higher values indicate more pronounced social anxiety symptoms during the last week.
Change in social anxiety; measured with the Social Interaction Anxiety Scale (SIAS) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The SIAS presents a widely used and well-validated questionnaire to assess social anxiety. It focuses on social interaction anxiety, a subdimension of social anxiety and consists of 20 five-point items (0 = "not at all", 1 = "a little", 2 = "quite", 3 = "strongly", 4 = "very strongly") with a value range extending from 0 to 80 with higher values indicating severer social interaction anxiety.
Imagination abilities; measured with the Spontaneous Use of Imagery Scale (SUIS) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The SUIS is used to assess the subject's ability to use mental images. This ability might be a requirement to profit from the reward training since it is partly based on imagination exercises. The training might also lead to an improvement in this ability by practicing them repeatedly in everyday life. The SUIS consists of 18 five-point items (1 = "always applies", 3 = "applies half the time", 5 = "never applies") which the test subject can use to assess their spontaneous use of imagery in everyday life. Value range extends from 18 to 90 with higher values indicating frequent spontaneous use of imagery.
Vividness of mental images; measured with the Plymouth Sensory Imagery Questionnaire (PSI-Q) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The PSI-Q is used to assess the vividness of created mental images. The ability to create vivid mental images might be a requirement to profit from the reward training since it is partly based on imagination exercises. The training might also lead to an improvement in this ability by practicing it repeatedly in everyday life. The PSI-Q contains seven areas of imaginable experiences (visual, auditive, olfactory, gustatory, touch, kinesthetic and emotional), each with three examples (21 items total) on the basis of which the subject can rate their imagery experience from "no image at all" to "As vivid as real life" using a visual analog scale. Higher values indicate higher vividness of imagery.
Changes in feeling gratitude; measured with the Gratitude Questionnaire-Five-German (GQ-5-G) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale consists of five statements on the topic of gratitude, which the test subject is asked to rate on a seven-point scale (1 = "do not agree at all", 2 = "do not agree", 3 = "tend to disagree", 4 = "partly, partly", 5 = "tend to agree", 6 = "agree", 7 = "completely agree") in terms of their own agreement. Value range extends from 5 to 35 with higher values indicating a higher degree of gratitude.
Changes in perseverative thinking; measured with the Perseverative Thinking Questionnaire (PTQ) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale consists of 15 five-point items (0 = "never", 1 = "rarely", 2 = "sometimes", 3 = "frequently", 4 = "almost always") with statements about repetitive core features negative thinking, unproductiveness of repetitive negative thinking and mental capacity captured by repetitive negative thinking. The subject is asked to indicate whether the described is often or seldom the case. Value range extends from 0 to 60 with higher values indicating a higher degree of repetitive negative thinking.
Changes in use of emotion regulation strategies; measured with the Emotion Regulation Questionnaire (ERQ) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale consists of 10 seven-point items (1 = "not true at all", 4 = "neutral", 7 = "abolutely right") about emotion regulation strategies (6 items on reappraisal and 4 items on suppression) and their degree of usage. Value range extends from 10 to 70 with higher values indicating more usage of the named emotion regulation strategy.
Changes in feeling overall relaxed (single self-composed visual analog scale item) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  Item asking "How relaxed do you feel at the moment?"; answer to be indicated using a visual analog scale (0-100) with the poles "not at all relaxed" to "completely relaxed"; higher value indicates more relaxation
Changes in feeling stressed; measured with the Perceived Stress Questionnaire (PSQ) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale assesses the current subjective overall stress using 20 four-point items (1 = "almost never", 2 = "sometimes", 3 = "frequently", 4 = "most of the time") about the frequency of stress symptoms during the last four weeks. The value range extends from 20 to 80 with higher values indicating higher perceived stress.
Changes in general well-being; measured with the Short Form-8 Health Survey (SF-8-HS) from baseline to completion and baseline to follow-up | Baseline, 2 weeks (completion of intervention) and 3 months
  The scale assesses health-related quality of life during the last four weeks on the basis of eight items about general health, health-related restrictions, health-related difficulties in performance of daily tasks, intensity of pain, amount of energy, degree of health-related restrictions in contact with family or friends, degree of anxiety/depression/irritability and job performance. Scale is either six- or five-point with higher values indicating poorer quality of life. Value range extends from 8 to 42.
Unwanted effects of the intervention/negative intervention outcomes; measured with the Inventory for balanced recording of negative effects of psychotherapy (INEP) | 3 months
  The INEP conducts negative effects of psychotherapy interventions on the basis of 21 items with which the test subject can indicate whether they feel better or worse in different areas after the intervention than they did before with regard to, for example feeling better or worse or having more conflicts than before (items 1-6 use 7-point scales from 3 (e.g. "better") to -3 (e.g. "worse"), items 7-21 use 4-point scales (0 = "does not apply at all", 1 = "applies to a certain extent", 2 = "partially true", 3 = "totally true") . The test subjects are also asked whether they attribute the changes to the interventions or to other circumstances (items 1-15) or to describe their experiences (item 16-21). The wording of the items was adjusted to meet the purpose of the app-based intervention.
EMA-measures during active participation (part 1) | Three times daily (morning, afternoon, evening; accompanying the exercises) over the course of 14 days
  Activities since the last beep (multiple choice item with 16 different options such as "work/school/studies", "household" or "hobbys"), Current mood (six seven-point bipolar items with visual analog scales to assess momentary valence ("content" and "well" and their respective opposites as poles of the scale), calmness ("calm" and "relaxed") and energetic arousal ("awake" and "full of energy")), Current symptoms of depression (two VAS-items on depressive symptoms (anhedonia and depressed mood); 0-100 with higher values indicating higher severity of current depressive symptoms), Current symptoms of (generalized) anxiety (two VAS-items on symptoms of anxiety (nervousness/anxiety/tension and not being able to control one's worry); 0-100 with higher values indicating higher severity of generalized anxiety symptoms), Current degree of rumination (VAS-item on repetitive thinking about a past event; 0-100 with higher values indicating higher degrees of rumination)
EMA-measures during active participation (part 2) | Three times daily (morning, afternoon, evening; accompanying the exercises) over he course of 14 days
  Current motivation to interact with other people (as a measure of motivated action; VAS-item; 0-100 with higher values indicating higher degrees of motivation), Current capacity of pleasure by interaction with other people (as a measure of consummatory pleasure; VAS-item; 0-100 with higher values indicating higher degrees of consummatory pleasure), Current capacity of pleasure by looking forward to interaction with other people (as a measure of anticipatory pleasure; VAS-item; 0-100 with higher values indicating higher degrees of anticipatory pleasure), Current expectation of pleasure by thinking about future interactions with other people (as a measure of anticipated pleasure; VAS-item; 0-100 with higher values indicating higher degrees of anticipated pleasure)
EMA-measures during active participation (part 3) | Three times daily (morning, afternoon, evening; accompanying the exercises) over the course of 14 days
  Current avoidance of interaction with other people (VAS-item; 0-100 with higher values indicating higher degrees of avoidance), Current mood directly before and after the training exercises (display of a smiley on the smartphone screen that reflects the subject's positioning of a VAS (0-100) from "very bad" to "very good" as a measure of the training exercise's effect on mood), Vividness of imagination (VAS-item (0-100) from "not at all vivid" to "very vivid" to assess the subject's imagination experience; item only used in the reward training condition), Positive emotions as produced by the training exercise (open text item; the subject is supposed to name all distinct positive emotions that came up in reaction to the exercise; item used in reward and relaxation condition)

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps-University Marburg, Marburg, Hesse, Germany